CLINICAL TRIAL: NCT02219724
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of MOXR0916 Administered Intravenously as a Single Agent to Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study to Assess Safety and Pharmacokinetics of MOXR0916 in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29313; 2014-001474-34 (EudraCT Number)
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- MOXR0916: Dose Escalation Stage (Experimental): Participants in different cohorts (according to MOXR0916 dose received) will receive escalating doses of MOXR0916 to determine the MTD or maximum administered dose (MAD) for 21 to 42 days.
  Interventions: Drug: MOXR0916
- MOXR0916: Expansion Stage (Experimental): Participants in different cohorts (according to different cancer types, prior therapy and mandatory procedures on study) will receive MOXR0916 at the highest dose level that has already been deemed to be tolerable in the dose escalation stage until disease progression, loss of clinical benefit or unacceptable toxicity, whichever occurred first (approximately up to 3 years).
  Interventions: Drug: MOXR0916

INTERVENTIONS:
Drug: MOXR0916 — MOXR0916 will be administered as intravenous infusion on Day 1 of each 21-day cycle.

SUMMARY:
This is a first-in-human, Phase 1, open-label, multicenter, dose-escalation study designed to evaluate the safety, tolerability, and pharmacokinetics of MOXR0916 administered intravenously in participants with locally advanced or metastatic solid tumors that have progressed after all available standard therapy or for which standard therapy has proven to be ineffective or intolerable, or is considered inappropriate. This study will consist of a screening period, an initial treatment period, a re-treatment period (for participants who discontinue MOXR0916 after demonstration of prolonged clinical benefit), and a post-treatment follow-up period. Participants will be enrolled in two stages: a dose-escalation stage and an expansion stage. The planned duration of the study is approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of locally advanced, recurrent or metastatic incurable solid malignancy that has progressed after all available standard therapy or for which standard therapy has proven to be ineffective or intolerable, or is considered inappropriate
* Confirmed availability of representative tumor specimens in paraffin blocks/unstained slides
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and end organ function
* For female participants of childbearing potential, agreement to use highly effective form(s) of contraception and to continue its use for 6 months after the last dose of MOXR0916

Exclusion Criteria:

* Any anti-cancer therapy, including chemotherapy, hormonal therapy, or radiotherapy, within 3 weeks prior to initiation of study treatment (hormonal therapy with gonadotropin-releasing hormone agonists or antagonists for prostate cancer and palliative radiotherapy greater than (>) 2 weeks prior to Cycle 1, Day 1 are allowed)
* Eligibility based on prior treatment with immunomodulatory agents depends on the mechanistic class of the drug and the cohort for which the participant is being considered
* Adverse events from prior anti-cancer therapy that have not resolved to Grade less than or equal to (</=) 1 except for alopecia or endocrinopathy managed with replacement therapy
* Primary central nervous system (CNS) malignancy, or untreated/active CNS metastases
* Leptomeningeal disease
* Malignancies other than disease under study within 5 years
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus infection
* Active hepatitis B or active hepatitis C
* Severe infections within 4 weeks or signs or symptoms of infection within 2 weeks prior to Cycle 1
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Significant cardiovascular disease
* Known clinically significant liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2019-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities (DLTs) | Day 1 Up to Day 21 or 42
Percentage of Participants With Adverse Events (AEs) by Severity as Graded per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) | Baseline up to 90 days after the last dose of study treatment, or until the initiation of another systemic anti-cancer therapy, whichever occurs first (approximately up to 3 years)

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MOXR0916 | Baseline up to 21 to 42 days
Recommended Phase II Dose of MOXR0916 | Baseline up to 21 to 42 days
Percentage of Participants With Anti-MOXR0916 Antibodies | Pre-dose (Hour [Hr] 0) on Day (D) 1 of Cycles (Cy) 1,2,3,4,8,12,16, & then every 8 Cy up to treatment discontinuation visit (TDV) (up to approximately 3 years) (1 Cy=21 days), thereafter every 30 days for up to 120 days after treatment discontinuation
Number of Cycles of MOXR0916 Treatment Received | Baseline up to approximately 3 years
Mean MOXR0916 Dose Administered During Study | Baseline up to approximately 3 years
Area Under the Serum Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) of MOXR0916 | Cy1 (1Cy=21 days): Predose (Hr0), 0.5,24,72 hrs postinfusion (infusion duration=1.5 hrs) on D1; on D8, 15; Cy2-7: Hr0, 0.5 hrs postinfusion on D1; Cy8,12,16, then every 8 Cy up to TDV (approx. 3 years): Hr0 on D1; every 30 days after TDV up to 120 days
Maximum Observed Serum Concentration (Cmax) of MOXR0916 | Cy1 (1Cy=21 days): Predose (Hr0), 0.5,24,72 hrs postinfusion (infusion duration=1.5 hrs) on D1; on D8, 15; Cy2-7: Hr0, 0.5 hrs postinfusion on D1; Cy8,12,16, then every 8 Cy up to TDV (approx. 3 years): Hr0 on D1; every 30 days after TDV up to 120 days
Minimum Observed Serum Concentration (Cmin) of MOXR0916 | Cy1 (1Cy=21 days): Predose (Hr0), 0.5,24,72 hrs postinfusion (infusion duration=1.5 hrs) on D1; on D8, 15; Cy2-7: Hr0, 0.5 hrs postinfusion on D1; Cy8,12,16, then every 8 Cy up to TDV (approx. 3 years): Hr0 on D1; every 30 days after TDV up to 120 days
Serum Clearance (CL/F) of MOXR0916 | Cy1 (1Cy=21 days): Predose (Hr0), 0.5,24,72 hrs postinfusion (infusion duration=1.5 hrs) on D1; on D8, 15; Cy2-7: Hr0, 0.5 hrs postinfusion on D1; Cy8,12,16, then every 8 Cy up to TDV (approx. 3 years): Hr0 on D1; every 30 days after TDV up to 120 days
Apparent Volume of Distribution at Steady State (Vss) of MOXR0916 | Cy1 (1Cy=21 days): Predose (Hr0), 0.5,24,72 hrs postinfusion (infusion duration=1.5 hrs) on D1; on D8, 15; Cy2-7: Hr0, 0.5 hrs postinfusion on D1; Cy8,12,16, then every 8 Cy up to TDV (approx. 3 years): Hr0 on D1; every 30 days after TDV up to 120 days
Percentage of Participants With Objective Response as Determined Using Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
Duration of Objective Response (DOR) as Determined Using RECIST v1.1 | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
Progression-free Survival (PFS) as Determined Using RECIST v1.1 | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
Percentage of Participants With Objective Response as Determined Using Modified RECIST | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
DOR as Determined Using Modified RECIST | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
PFS as Determined Using Modified RECIST | Baseline, end of Cycles 2, 4, 6, 8, and every 4 cycles thereafter (cycle length=21 days) until disease progression, death, another anti-cancer therapy initiation, loss to follow-up, consent withdrawal, or study termination (approximately up to 3 years)
Overall Survival (OS) | Baseline until death, loss to follow-up, withdrawal of consent, or study termination by the Sponsor (approximately up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (31):
- United States (12):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - University of Colorado, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - University Of Chicago Medical Center; Section Of Hematology/Oncology, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
  - Sint Augustinus Wilrijk, Wilrijk
- Canada (5):
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Yonsei University Health System/Severance Hospital, Seoul
- Spain (4):
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hosp de Madrid Norte Sanchinarro; Centro Integral; Onco Clara Campal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia